CLINICAL TRIAL: NCT06398171
Title: Exercise-induced Hypoalgesia in Patients With Knee Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Luis Suso, PhD, Cardenal Herrera University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EIH1
Record Dates: First submitted 2024-04-23; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Participants will perform 8 sessions of 4 sets of knee extension exercises during 1 month

SUMMARY:
The main objective of this study is to evaluate the differences in the phenomenon of exercise-induced hypoalgesia in patients with osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with severe knee OA (according to the clinical and radiographic criteria of the American College of Rheumatology Guidelines)

Exclusion Criteria:

* pain in the contralateral (non-studied) limb (maximum ≥80 of 100 mm on a visual analog scale (VAS) during daily activities),
* undergone another hip or knee joint replacement in the previous year
* any medical condition in which exercise was contraindicated

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Algometry | Before and after exercise (1 month)
  Pressure pain thresholds will be measured at the affected knee, the contralateral knee and the contralateral epicondyle.

IPD SHARING:
Plan to Share IPD: Undecided